CLINICAL TRIAL: NCT02207946
Title: Prospective, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of the Efficacy and Safety of NT 201 in the Unilateral Treatment of Essential Tremor of the Upper Limb
Brief Title: Botulinum Toxin A to Treat Arm Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ60201_2094_1
Record Dates: First submitted 2014-08-01; First posted 2014-08-04 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Essential Tremor of the Upper Limbs
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 200 Units incobotulinumtoxinA (Xeomin) (Experimental): Single injection cycle, total dose of up to 200 Units, intramuscular injection into muscles of wrist (mandatory) and shoulder and/or elbow (both optional).
  Interventions: Drug: IncobotulinumtoxinA
- Placebo (Placebo Comparator): Single injection cycle, intramuscular injection into muscles of wrist (mandatory) and shoulder and/or elbow (both optional).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IncobotulinumtoxinA — Active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl).
  Other Names: Xeomin; NT 201; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
  Arms: 200 Units incobotulinumtoxinA (Xeomin)
Drug: Placebo — Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl).
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the efficacy and safety of a single, kinematic-analysis-based intramuscular injection of NT 201, compared with placebo, in moderate to marked essential tremor of the upper limb.

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosis of 'definite essential tremor' in accordance with modified TRIG criteria, as follows:

  * Bilateral postural tremor with or without kinetic tremor, involving hands and forearms, that is visible and persistent.
  * It is to be noted that:
  * Tremor of other body parts may be present in addition to upper limb tremor.
  * Bilateral tremor may be asymmetric.
  * Tremor is reported by patient to be persistent, although the amplitude may fluctuate.
* First onset of essential tremor at least 6 months before screening with stability of the tremor symptoms over 4 weeks and in the opinion of the investigator definite diagnosis of essential tremor.
* Moderate-to-marked upper-limb postural and/or kinetic tremor at wrist level, corresponding to Fahn-Tolosa-Marin upper-limb tremor rating of at least 2 categories (scale part C, items 16-23) in the limb to be treated between of 2 or higher.
* Visible tremor at wrist level in at least one of the four positions/tasks used in kinematic assessments
* Tremor deemed by the investigator to require a treatment with 30 - 200 U NT 201 for a treatment of up to three joints of the selected upper limb (wrist treatment mandatory).
* Stable concomitant anti-tremor medication and no clinically relevant findings in routine laboratory examinations.

Main Exclusion Criteria:

* Any neurological signs abnormal for the subject's age, other than the tremor itself and Froment's maneuver.
* Exposure to the following tremorogenic drugs: Lithium, Valproic acid, Amiodarone, typical and atypical neuroleptics. Exposure to other than the listed tremorogenic or potentially tremorogenic drugs is allowed only if, in the opinion of the investigator, this will not interfere with the study drug evaluation. In these cases, a stable medication should be reached 4 weeks before screening and intended for the time during the study drug evaluation.
* Trauma to the central nervous system or the nerves of the target limb within the three months preceding the onset of tremor.
* Evidence of psychogenic origins of tremor.
* Life habits (e.g. smoking, alcohol or substance abuse) prejudicial to study participation.
* Prior surgery to treat tremor
* Recent (16 weeks) treatment with any Botulinum toxin product for any reason.
* Relevant recent or planned surgery or other specified relevant treatments and/or concomitant disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12-05 (Actual); Primary Completion 2016-05-09 (Actual); Study Completion 2016-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (6):
- Merz Investigational Site #0010191, New York, New York, United States
- Canada (5):
  - Merz Investigational Site #0010317, Winnipeg, Manitoba
  - Merz Investigational Site #0010089, Halifax, Nova Scotia
  - Merz Investigational Site #0010078, Toronto, Ontario
  - Merz Investigational Site #0010305/1, Toronto, Ontario
  - Merz Investigational Site #0010305/2, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jog M, Lee J, Scheschonka A, Chen R, Ismail F, Boulias C, Hobson D, King D, Althaus M, Simon O, Dersch H, Frucht S, Simpson DM. Tolerability and Efficacy of Customized IncobotulinumtoxinA Injections for Essential Tremor: A Randomized, Double-Blind, Placebo-Controlled Study. Toxins (Basel). 2020 Dec 20;12(12):807. doi: 10.3390/toxins12120807. PMID 33419261

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The multicenter study was conducted at 6 investigational sites in the United States and Canada.
Pre-assignment Details: A total of 52 participants were screened, out of which 30 participants were randomized and treated.
Groups:
- IncobotulinumtoxinA 30 to 200 Units: Participants received incobotulinumtoxinA (also known as NT 201) between 30 to 200 units (U), powder for solution for injection, intramuscular injection, unilaterally into the muscles of the wrist, and optionally, into the elbow and shoulder as based upon kinematic analysis, in a single injection session on Day 1 (Visit 2). The maximum dose per injection site (more than one site per muscle were possible) was 25 U incobotulinumtoxinA.
- Placebo: Participants received placebo solution matched to the volume of incobotulinumtoxinA solution, intramuscular injection, unilaterally into the muscles of the wrist, and optionally, into the elbow and shoulder as based upon kinematic analysis, in a single injection session on Day 1 (Visit 2). The maximum dose per injection site (more than one site per muscle were possible) was 25 U incobotulinumtoxinA placebo.
Period: Overall Study
Arm/Group | IncobotulinumtoxinA 30 to 200 Units | Placebo
Started | 19 | 11
Completed | 18 | 10
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety evaluation set (SES) was the subset of all participants who received study medication (incobotulinumtoxinA or placebo) at least once.
Groups:
- IncobotulinumtoxinA 30 to 200 U: Participants received incobotulinumtoxinA (also known as NT 201) between 30 to 200 U, powder for solution for injection, intramuscular injection, unilaterally into the muscles of the wrist, and optionally, into the elbow and shoulder as based upon kinematic analysis, in a single injection session on Day 1 (Visit 2). The maximum dose per injection site (more than one site per muscle were possible) was 25 U incobotulinumtoxinA.
- Total: Total of all reporting groups
Arm/Group | IncobotulinumtoxinA 30 to 200 U | Placebo | Total
Number analyzed (Participants) | 19 | 11 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (10.6) | 68.2 (10.2) | 68.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 9 | 6 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 11 | 28
  Black or African American | 1 | 0 | 1
  Asian | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in Maximum Angular Tremor Amplitude of the Wrist (Injected Limb)
Description: No primary efficacy variables are defined for this study. One of the secondary outcome measures is used for CTgov protocol registration and results reporting purposes only. TremorTek is a tremor kinematic analytics investigational device which is used to measure maximum angular tremor amplitude at wrist of the injected limb (unit: degrees). Angular tremor amplitude is the measure of tremor severity. Reduction of angular tremor amplitude at wrist of the injected limb represents tremor improvement.
Time Frame: Baseline up to Week 4
Population: The full analysis set (FAS) was defined as the subset of participants who received study medication (incobotulinumtoxinA or placebo) at least once, and for whom a post-baseline value of any efficacy variable was measured.
Measure: Mean (Standard Deviation); unit: degree
Groups:
- IncobotulinumtoxinA 30 to 200 U: Participants received incobotulinumtoxinA (also known as NT 201) between 30 to 200 units (U), powder for solution for injection, intramuscular injection, unilaterally into the muscles of the wrist, and optionally, into the elbow and shoulder as based upon kinematic analysis, in a single injection session on Day 1 (Visit 2). The maximum dose per injection site (more than one site per muscle were possible) was 25 U incobotulinumtoxinA.
Arm/Group | IncobotulinumtoxinA 30 to 200 U | Placebo
Number analyzed (Participants) | 18 | 11
degree | -0.47 (0.63) | 0.07 (0.88)
Statistical Analysis 1: Comparison: IncobotulinumtoxinA 30 to 200 U vs Placebo; Least square (LS) means are from analysis of covariance (ANCOVA) with treatment and site included as fixed factors and baseline included as covariate; Test type: Superiority; p = 0.144, ANCOVA; LS mean difference = -0.43, 95% CI 2-sided [-1.02 to 0.16], Standard Error of Mean 0.28

2. Secondary Outcome: Change From Baseline to Week 4 in Maximum Log-transformed Accelerometric Tremor Amplitude at Wrist Level (Injected Limb)
Description: TremorTek is a tremor kinematic analytics investigational device which is used to measure maximum log-transformed accelerometric tremor amplitude at wrist level of the injected limb (unit: meter per square second [m/s˄2]). Log-transformed accelerometric tremor amplitude is a measure of tremor severity reflecting the non-vectoral intensity of tremor. Reduction of log-transformed accelerometric tremor amplitude at wrist level of the injected limb represents a tremor improvement.
Time Frame: Baseline up to Week 4
Population: The FAS was defined as the subset of participants who received study medication (incobotulinumtoxinA or placebo) at least once, and for whom a post-baseline value of any efficacy variable was measured.
Measure: Mean (Standard Deviation); unit: log[m/s˄2]
Arm/Group | IncobotulinumtoxinA 30 to 200 U | Placebo
Number analyzed (Participants) | 18 | 11
log[m/s˄2] | -0.73 (0.63) | 0.05 (0.38)

3. Secondary Outcome: Change From Baseline to Week 4 in Fahn-Tolosa-Marin (FTM) Tremor Score in Injected Limb (Item 5 [Right Upper Extremity] or 6 [Left Upper Extremity])
Description: The FTM tremor rating scale is used for evaluation of tremor severity and function and consists of three parts (A, B, C). For this outcome measure the score of FTM scale item 5 ("right upper extremity") or item 6 ("left upper extremity") is used (both items are from part A). The outcome values are calculated as the sum of the three functions "at rest", "with posture holding", and "with action and intention". The score for each item ranges from 0 (normal) to 4 (severe), that is, the possible values range from 0 to 12.
Time Frame: Baseline up to Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IncobotulinumtoxinA 30 to 200 U | Placebo
Number analyzed (Participants) | 18 | 11
score on a scale | -1.9 (1.9) | -0.5 (1.8)

4. Secondary Outcome: Change From Baseline to Week 4 in FTM Motor Performance Score (Items 11-15)
Description: The FTM tremor rating scale was used for evaluation of tremor severity and function. This investigator-assessed scale consists of 3 parts (A, B and C). Part A: Tremor location/Severity rating (items 1-10); Part B: Specific motor tasks / Function rating (items 11-15). Ratings for five motor tasks (handwriting, drawing [large/small spiral, line], and pouring); and Part C: Functional disabilities resulting from tremor/activities of daily living (items 16-23). For this outcome measure, the sum of the five FTM motor performance items (from Part B) were used: item 11 ('handwriting for dominant hand only' - irrespective of its injection or non-injection), items 12 to 15 ('drawing large and small spiral', 'line drawing', 'pouring' for the injected upper limb). The score for each item ranges from 0 (normal) to 4 (severe). Possible values range for total FTM motor performance score: 0-20.
Time Frame: Baseline up to Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IncobotulinumtoxinA 30 to 200 U | Placebo
Number analyzed (Participants) | 18 | 11
score on a scale | -2.8 (1.6) | -0.8 (2.0)

5. Secondary Outcome: Participant's Global Impression of Change Scale (GICS) at Week 4
Description: The GICS was used to measure the participant's impression of change due to treatment. The response option was a common 7-point Likert scale, with the following values: +3 (very much improved); +2 (much improved); +1 (minimally improved); 0 (no change); -1 (minimally worse); -2 (much worse); -3 (very much worse).
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IncobotulinumtoxinA 30 to 200 U | Placebo
Number analyzed (Participants) | 18 | 11
score on a scale | 0.6 (0.6) | 0.3 (0.6)

6. Secondary Outcome: Investigator's Global Impression of Change Scale (GICS) at Week 4
Description: The GICS was used to measure the investigator's impression of change due to treatment. The response option was a common 7-point Likert scale, with the following values: +3 (very much improved); +2 (much improved); +1 (minimally improved); 0 (no change); -1 (minimally worse); -2 (much worse); -3 (very much worse).
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IncobotulinumtoxinA 30 to 200 U | Placebo
Number analyzed (Participants) | 18 | 11
score on a scale | 0.8 (0.7) | 0.1 (0.7)

ADVERSE EVENTS:
Time Frame: From screening up to Week 24
Description: The investigator asked the participant for adverse events (AEs) systematically at each visit.
Arm/Group | IncobotulinumtoxinA 30 to 200 U | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/19 | 2/11
Other Adverse Events (participants affected / at risk) | 9/19 | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IncobotulinumtoxinA 30 to 200 U (N=19) | Placebo (N=11)
Influenza like illness (General disorders) | 0 | 1
Chest discomfort (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IncobotulinumtoxinA 30 to 200 U (N=19) | Placebo (N=11)
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Cystitis (Infections and infestations) | 1 | 0
Eyelid infection (Infections and infestations) | 1 | 0
Genital infection (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Injection site bruising (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.